CLINICAL TRIAL: NCT00057967
Title: Phase II Trial Of Campath-1H In Patients With Relapsed/Refractory Advanced Mycosis Fungoides or Sezary Syndrome
Brief Title: Alemtuzumab in Treating Patients With Relapsed or Refractory Advanced Mycosis Fungoides or Sézary Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 99H8; NU 99H8 (Other: Northwestern University); STU00012258 (Other: Northwestern University IRB)
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-01

CONDITIONS: Lymphoma
Keywords: recurrent mycosis fungoides/Sezary syndrome; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment arm (Experimental): alemtuzumab
  Interventions: Biological: alemtuzumab

INTERVENTIONS:
Biological: alemtuzumab — Will be administered as a two-hour IV infusion with a target dose of 30 milligrams three times a week for a maximum of 12 weeks.
  Other Names: Campath; MabCampath; Campath-1H

SUMMARY:
RATIONALE: Monoclonal antibodies such as alemtuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: This phase II trial is studying how well alemtuzumab works in treating patients with relapsed or refractory advanced mycosis fungoides or Sézary syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients with relapsed or recurrent advanced mycosis fungoides or Sézary syndrome treated with alemtuzumab.
* Determine the toxicity of this drug in these patients.

OUTLINE: Patients receive alemtuzumab IV over 2 hours three times per week. Treatment continues for up to 12 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed mycosis fungoides or Sézary syndrome

  * Stage IB-IVB
* Measurable disease

  * One or more indicator lesions
  * No prior radiotherapy to areas of measurable disease unless there is clear disease progression at the site or measurable disease outside the area of prior radiotherapy
  * Generalized erythrodermia patients with evaluable disease only are allowed
* Must have failed at least 1 prior systemic therapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* WHO 0-2

Life expectancy

* At least 3 months

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 2.2 mg/dL
* AST or ALT no greater than 2 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2 times ULN

Renal

* Creatinine no greater than 2.0 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No acute infection requiring intravenous antibiotics
* No other prior neoplasm except treated squamous cell or basal cell skin cancer, treated carcinoma in situ of the cervix, or other cancer that received surgical treatment only from which patient has been disease free for at least 5 years

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior biologic therapy

Chemotherapy

* More than 4 weeks since prior chemotherapy

Endocrine therapy

* More than 4 weeks since prior topical steroids

Radiotherapy

* See Disease Characteristics
* At least 2 weeks since prior radiotherapy (local control or palliative)
* No concurrent radiotherapy to any lesion

Surgery

* Recovered from prior major surgery

Other

* Recovered from prior therapy
* No other concurrent proven or investigational antineoplastic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2000-07; Primary Completion 2007-06-26 (Actual); Study Completion 2010-07-26 (Actual)

PRIMARY OUTCOMES:
Determine response rate associated with Campath-1H therapy in patients with relapsed Mycosis Fungoides/Sezary Syndrome | At baseline, weekly while on treatment, then once when patient goes off study
  Response rate associated with Campath-1H therapy in patients with relapsed Mycosis Fungoides/Sezary Syndrome will be assessed by medical photograph (skin lesion) measurements or by CT scan for internal lesions upon study entry, weekly while on study, then once when patient goes off study
Collect data on toxicity associated with Campath-1H therapy | At baseline and then every 2 weeks while on therapy
  Toxicity of this drug will be assessed upon study entry and then every 2 weeks while on therapy by blood tests

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M. Kuzel, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois